CLINICAL TRIAL: NCT05747989
Title: A Comparison of Tissue Adhesive Material and Suture as Wound-closure Techniques
Brief Title: A Comparison of Tissue Adhesive Material and Suture as Wound-closure Techniques Following Carpal Tunnel Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Vedran Kovacic, Clinical Professor, Head of Internal Division ICU, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500-03/22-01/41
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin stitched with two-component skin adhesive (Active Comparator): After subcutaneous stitches a two-component skin adhesive, Glubran Tiss 2®, will be applied. G Each subject will receive 0.35 mL of Glubran Tiss® in the open wound, and before bandaging, subjects rested for 20 minutes for a polymerization process.
  Interventions: Procedure: two-component skin adhesive, Glubran Tiss 2
- skin stitched with transcutaneous nylon sutures (Placebo Comparator): The skin is stitched with transcutaneous nylon sutures (polypropylene-polyethylene monofilament, non-absorbable surgical suture) 4-0. (Optilene® DSMP 19, 3/8 needle, thread size 4/0
  Interventions: Procedure: skin is stitched with transcutaneous nylon sutures

INTERVENTIONS:
Procedure: two-component skin adhesive, Glubran Tiss 2 — After subcutaneous stitches a two-component skin adhesive, Glubran Tiss 2®, will be applied. G Each subject will receive 0.35 mL of Glubran Tiss® in the open wound, and before bandaging, subjects rested for 20 minutes for a polymerization process.
  Arms: skin stitched with two-component skin adhesive
Procedure: skin is stitched with transcutaneous nylon sutures — The skin is stitched with transcutaneous nylon sutures (polypropylene-polyethylene monofilament, non-absorbable surgical suture) 4-0
  Arms: skin stitched with transcutaneous nylon sutures

SUMMARY:
Participants will be randomly assigned to suture-based wound closure (n=50) or tissue adhesive-based wound closure (n=50) with two-component skin adhesive Glubran Tiss 2®. The outcomes will be assessed during the follow-up period at intervals of 2, 6, and 12 weeks postoperatively. A scar assessment will be using the POSAS (Patient and Observer Scar Assessment Scale) and cosmetic VAS (Visual Analog Scale). The VNRS (Verbal Number Rating Scale) will used to assess pain.

ELIGIBILITY:
Inclusion Criteria: (all of the above)

* age >18 years
* carpal tunnel syndrome
* weakness of thumb abduction
* with atrophy of the thenar
* median nerve conduction impairment estimated by electromyography

Exclusion Criteria: (one or more)

* threatening haemorrhagic complications (patients with peroral anticoagulation and/or antithrombotic therapy)
* previous wrist trauma or surgery on the wrist region
* another aetiology of neuropathy
* previous allergic reactions (with lidocaine, cyanoacrylate, formaldehyde, tapes, or adhesives)
* personal or family history of keloids or hypertrophic scars
* severe general illness with cachexia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 12 weeks
  scar assessment
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6

SECONDARY OUTCOMES:
Verbal Number Rating Scale (VNRS) - to assess the degree of pain | 12 weeks
  degree of pain
  A Verbal Number Rating Scale (VNRS) was used to assess the degree of pain in the hand before and the day after surgery, as well as at 2, 6, and 12-week intervals during the follow-up period. The VNRS is a verbal self-report instrument with a 0 - 10 numeric rating scale, where 0 represents no pain and 10 represents the most severe pain possible
VAS - Visual Analog Scale | 12 weeks
  scar assessment
  VAS (Visual Analog Scale) assessment form was filled out by the patient at the 2, 6, and 12-week intervals. The cosmetic-VAS is a 0-100 scale with "worst scar" written at the left end (0) and "best scar" written at the right end (100)

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Kovacic, Prof, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University Hospital of Split, 21000 Croatia, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available on request.